CLINICAL TRIAL: NCT04618315
Title: Patient-Centered Hearing Aid Trial: Comparison of Direct to Consumer Delivery Models for Hearing Devices
Brief Title: P-CHAT: Comparison of Direct to Consumer Delivery Models for Hearing Devices
Acronym: P-CHAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Sumit Dhar, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HL-2019C1-16094
Record Dates: First submitted 2020-10-31; First posted 2020-11-05 (Actual); Results first posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Hearing Aids; Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Intervention Model Description: Three arm blinded randomized control trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The principle investigators and the audiologists conducting the outcome measures will be blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Audiology-Based Best Practice (Active Comparator): Hearing aids will be fit using current best practices used by audiologists to fit hearing aids.
  Interventions: Device: Hearing Aids
- Consumer Decides (Experimental): Hearing aids will be self fit by patients using an interactive application on a tablet computer. Patients will choose their preferred hearing aid settings after comparing four settings with varying loudness levels.
  Interventions: Device: Hearing Aids
- Efficient Fitting (Experimental): Hearing aids will be self fit by patients using an interactive application on a tablet computer. Patients will choose their preferred hearing aid settings after comparing four settings with varying base and treble settings.
  Interventions: Device: Hearing Aids

INTERVENTIONS:
Device: Hearing Aids — Receiver-in-the-ear hearing aids.

SUMMARY:
Satisfaction and benefit from hearing aids fit using two patient self fit methods will be compared against those fit using audiology-based best practices. Individuals between the ages of 50 and 79 years of age will be randomly assigned to one of three fitting methods. Benefit and satisfaction will be evaluated six weeks and six months after the initial fitting.

DETAILED DESCRIPTION:
Hearing aids are the most pertinent treatment for most adults with hearing loss, a pervasive chronic health problem in ~40% of those over the age of 60 years. Only 20% of these individuals purchase and use hearing aids. The Over-the-Counter Hearing Aid Act of 2017 is designed to increase affordability and accessibility, and thereby adoption, of hearing aids. While this legislation directs the Food and Drug Administration (FDA) to create and administer this new channel of hearing aid provision by 2020, best practices related to hearing aid provision without the involvement of a professional, licensed provider have not been explored and established. Patients do not have the evidence they need to decide between modes of acquiring hearing aids. The current proposal addresses the specific knowledge gap of efficacious direct-to-consumer hearing aid delivery models. Two methods of patient-driven methods of selecting and fitting hearing aids will be compared against audiology-based best practice fitting. Individuals who perceive mild or moderate hearing difficulty will be randomly assigned to one of three fitting arms. Satisfaction and benefit from hearing aids will be assessed at six weeks and six months after initial fit.

ELIGIBILITY:
Inclusion Criteria:

* 50 - 79 years old.
* Mild or moderate hearing difficulty.
* Normal cognition.
* No prior hearing aid experience.
* Ability and willingness to pay privately ($650.00) for hearing aids
* Ability to read and understand English
* Symmetric hearing loss, no greater than moderate in degree

Exclusion Criteria:

-

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sumitrajit Dhar, Principal Investigator — Northwestern University
Locations (4):
- United States (4):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Northwestern University Center for Audiology, Speech, Language, and Learning, Evanston, Illinois
  - Sertoma Speech and Hearing Center, Palos Hills, Illinois
  - University of Texas Medical Branch, Galveston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared at the Patient-Centered Outcomes Data Repository
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12 months after study completion through the PCORI data sharing platform.
Access Criteria: Requests will be evaluated first by PCODR staff who will then consult with PIs before approving access.

RESULTS

PARTICIPANT FLOW:
Period: 6-Week Primary Observation Point
Arm/Group | Audiology-Based Best Practice | Consumer Decides | Efficient Fitting
Started | 190 | 193 | 201
Completed | 182 | 172 | 178
Not Completed | 8 | 21 | 23
Period: 6-Month Secondary Observation Point
Arm/Group | Audiology-Based Best Practice | Consumer Decides | Efficient Fitting
Started | 182 | 172 | 178
Completed | 152 | 132 | 140
Not Completed | 30 | 40 | 38

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Audiology-Based Best Practice | Consumer Decides | Efficient Fitting | Total
Number analyzed (Participants) | 190 | 193 | 201 | 584
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.42 (6.95) | 69.81 (6.71) | 69.1 (6.71) | 69.11 (6.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 104 | 114 | 329
  Male | 79 | 89 | 87 | 255
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 4 | 15
  Not Hispanic or Latino | 184 | 188 | 197 | 569
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 1 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 2 | 7
  White | 176 | 187 | 192 | 555
  More than one race | 8 | 2 | 2 | 12
  Unknown or Not Reported | 0 | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 190 | 193 | 201 | 584
Better Ear 4-Frequency (0.5, 1, 2, 4 kHz) Pure Tone Average [Mean (Standard Deviation); unit: dB HL] | 32.1 (9.04) | 32.64 (9.21) | 31.47 (9.06) | 32.06 (9.1)
Montreal Cognitive Assessment [Mean (Standard Deviation); unit: units on a scale] — The Montreal Cognitive Assessment or MoCA is a screening test for cognitive function. The minimum and maximum scores possible are 0 and 30, respectively. The higher the score the better the cognitive function.
  units on a scale | 26.28 (1.93) | 26.18 (1.90) | 26.37 (1.96) | 26.28 (1.93)
Hearing Handicap Inventory - Global [Mean (Standard Deviation); unit: units on a scale] — The Hearing Handicap Inventory is a self-report of hearing difficulties in various situations. The scores can range between 0-100. A higher score indicates greater difficulty in hearing.
  units on a scale | 39.35 (18.83) | 39.66 (18.26) | 37.51 (19.37) | 38.82 (18.82)
Profile of Hearing Aid Performance/Benefit [Mean (Standard Deviation); unit: units on a scale] — The Profile of Hearing Aid Performance/Benefit is a self-report of performance with hearing aids. Two measures are obtained, one prior to hearing aid use and the second with hearing aids. The difference between the two scores is the benefit score that can range between 0-99. The higher the number the greater the perceived benefit with the hearing aids.
  units on a scale | 39.77 (14.21) | 40.05 (14.76) | 38.55 (14.86) | 39.44 (14.6)

OUTCOME MEASURES:

1. Primary Outcome: Profile of Hearing Aid Benefit
Description: 66-item self-assessment, disability-based inventory. Participants answer the questionnaire twice, first prior to use of hearing aids and then after hearing aid use. The questionnaire is scored between 0-99% with higher values representing greater difficulty. Benefit is reported as the difference between the two scores with a higher number signifying greater benefit.
Time Frame: 6 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Audiology-Based Best Practice | Consumer Decides | Efficient Fitting
Number analyzed (Participants) | 182 | 172 | 178
score on a scale | 23.34 [21.43 to 25.26] | 23.27 [21.54 to 25] | 23.33 [21.25 to 25.12]

2. Secondary Outcome: Hearing Handicap Inventory for the Elderly
Description: A self-administered scale to identify problems related to hearing loss. The questionnaire has 25 items and can be scored between 0 and 100. The score after hearing aid use is subtracted from the baseline score (prior to hearing aid use) to obtain the benefit score. The higher the difference the greater the benefit.
Time Frame: 6 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Audiology-Based Best Practice | Consumer Decides | Efficient Fitting
Number analyzed (Participants) | 182 | 172 | 178
score on a scale | 20.65 [18.11 to 23.19] | 21.83 [19.42 to 24.23] | 19.15 [16.59 to 21.73]

3. Other Pre Specified Outcome: Duration of Hearing Aid Use
Description: Average hours of hearing aid use per day.
Time Frame: 6 weeks
Measure: Mean (95% Confidence Interval); unit: hours/day
Arm/Group | Audiology-Based Best Practice | Consumer Decides | Efficient Fitting
Number analyzed (Participants) | 182 | 172 | 178
hours/day | 8.42 [7.91 to 8.92] | 7.18 [6.64 to 7.72] | 6.83 [6.32 to 7.34]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Audiology-Based Best Practice | Consumer Decides | Efficient Fitting
All-Cause Mortality (participants affected / at risk) | 0/182 | 0/172 | 0/178
Serious Adverse Events (participants affected / at risk) | 0/182 | 0/172 | 0/178
Other Adverse Events (participants affected / at risk) | 3/182 | 3/172 | 5/178
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Audiology-Based Best Practice (N=182) | Consumer Decides (N=172) | Efficient Fitting (N=178)
Receiver Dome in Ear (Ear and labyrinth disorders) | 2 (2) | 2 (2) | 4 (4) — The hearing aid receiver dome remained in the ear canal after the hearing aid was removed.
Ear Conditions (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 2 (2) — Complaints of ear pain, fullness, and/or itching
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) — Experience ringing in the ear
Reduced Hearing (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) — Complaint of reduced hearing ability

LIMITATIONS AND CAVEATS:
This study was initiated in 2020 before the approval of OTC hearing aids. Therefore, the devices used may not represent the quality of OTC hearing aids at any given time. The fitting methods used were derived from previous validation studies by the investigators. These results may not be valid for all self-fitting methods used in OTC hearing aids. Finally, the participants enrolled may not represent the demographic distribution of the United States or the areas in which the study was conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-10-04): https://cdn.clinicaltrials.gov/large-docs/15/NCT04618315/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-18): https://cdn.clinicaltrials.gov/large-docs/15/NCT04618315/SAP_002.pdf